CLINICAL TRIAL: NCT03272594
Title: The Influence of Breastfeeding on Pain-specific Event-related Potentials and Bio-behavioural Indicators of Procedural Pain in Newborns: A Randomized Controlled Trial
Brief Title: The Influence of Breastfeeding on Cortical Activity During Procedures
Acronym: iCAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Britney Benoit (Other)
Collaborators: Dalhousie University (Other); IWK Health Centre (Other)
Responsible Party: Sponsor-Investigator, Britney Benoit, Doctoral Candidate, Dalhousie University School of Nursing, IWK Health Centre
Organization: IWK Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1021795
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Pain; Neonatal
Keywords: Neonatal pain; Pediatric pain; Pain assessment; Breastfeeding; Sucrose; Randomized controlled trial; Behavioural pain response; Neurophysiological pain response
MeSH Terms: conditions — Pain; Breast Feeding | interventions — Lactation; Sucrose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two research assistants (RA1, RA2) who are blinded to the intervention condition will be hired to complete facial coding and calculation of infant PIPP-R scores. Each research assistant will only code data for infants in the breastfeeding condition (RA1) or the sucrose condition (RA2) and will not be aware of whether they are watching infant responses to noxious or non-noxious stimulation. To minimize observer bias, research assistants will not be informed of the study design, will not be permitted to attend data collection sessions, and will not share datasets or communicate with the other research assistant regarding the study. During data collection, up close video recording of only the infants face will be completed to attempt to keep coders blind to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breastfeeding (Experimental)
  Interventions: Other: Breastfeeding
- 24% oral sucrose (Active Comparator)
  Interventions: Drug: 24% oral sucrose

INTERVENTIONS:
Other: Breastfeeding — Infants will be placed in skin-to-skin contact with their mother at least five minutes prior to heel lance to allow time to settle and initiate breastfeeding. Breastfeeding position will be determined based on individual maternal preference in order to optimize feeding as well as to facilitate ease of access to the infant's foot for blood collection, while also attempting to minimize disruption of continuous EEG, heart rate, oxygen saturation, and video recording. Active breastfeeding will be facilitated to ensure it takes place for a minimum of two minutes prior to heel lance, and will continue until the procedure is completed.
  Arms: Breastfeeding
Drug: 24% oral sucrose — Administration of 24 percent oral sucrose will occur two minutes prior to the heel lance. Non-nutritive sucking will be offered using a gloved finger or pacifier (based on parental preference) immediately following administration of the complete 24 percent oral sucrose dose.
  Arms: 24% oral sucrose

SUMMARY:
Background: Even the healthiest infants undergo painful procedures as part of universal medical care. Untreated early pain is associated with heightened pain response during later procedures in infancy and alteration in response to pain in childhood. Oral sucrose is currently considered the standard of care for acute pain relief in infants. Compelling evidence from 57 randomized controlled trials suggests that oral sucrose reduces bio-behavioral pain response. However, recent data examining the influence of oral sucrose on pain-specific brain activity measured using electroencephalogram (EEG) questions the efficacy of this intervention for reducing pain in the infant brain. Evidence supports the effectiveness of breastfeeding as a pain relieving intervention, however, no studies to date have examined the effect of breastfeeding on pain-specific activity in the newborn brain.

Aims: The primary aim of this study is to examine the influence of breastfeeding in comparison to oral sucrose on pain-specific activity in the newborn brain during a heel lance. The secondary aim will be to determine if there is convergence among outcome measures in either of the intervention conditions.

Methods: Utilizing a single blind, randomized controlled trial design, 126 healthy term infants will be recruited within the first two days of life. Infants will be randomized to have a medically indicated heel lance completed in one of two possible conditions: 1) breastfeeding (n = 63) or 2) sucrose in an infant cot (n = 63). Infants will not be eligible for study participation if they show signs of lower limb tissue damage, have had previous surgery or intraventricular hemorrhage, are born to opioid using mothers or with significant genetic disorders, are unable to breastfeed, or have contraindications to sucrose administration. Pain-specific brain activity will be recorded on EEG for the duration of the blood collection. Infant facial response will be video recorded, and heart rate and oxygen saturation will be measured for calculation of Premature Infant Pain Profile-Revised (PIPP-R) Score, a reliable and valid bio-behavioral measure of pain in infants' 26-44 weeks gestational age. For infants randomized to the breastfeeding condition, data collection will begin with recording of a one-minute baseline (BL1). Following this, a non-painful control stimulus will be applied to the infant's foot to capture a baseline response on EEG to a non-painful event. The infant will then be transferred to the mother and active breastfeeding will be facilitated. A second baseline (BL2) will be recorded prior to heel lance. Pain response will be recorded from the initiation of the heel lance until procedure completion. In the sucrose condition, all monitoring will take place while the infant is in a cot (considered standard of care). Procedures will be consistent with those outlined above with the exception of administration of 24% oral sucrose two minutes prior to the heel lance. Analysis and inference will be calculated based on the intention-to-treat principle. Data from the EEG recording will be grouped into basic waveforms using principal component analysis. Two one-way analysis of variances will be used to assess the effect of stimulation type (non-painful control, painful heel lance) and treatment (24% oral sucrose, breastfeeding) on the principal components. To assess for the effect of treatment on PIPP-R score, group means will be compared using unpaired Student's t-tests.

Hypotheses: Infants in the breastfeeding condition will demonstrate both lower pain-specific brain response and lower bio-behavioral pain scores than infants in the sucrose condition.

Significance: This will be the first study to examine the effect of breastfeeding on pain-specific brain response in infants. In light of the negative consequences of unmanaged pain in infants, it is imperative that effective pain relieving interventions are utilized. Given recent evidence questioning the analgesic properties of sucrose, findings will have important implications for informing optimal pain management practices in infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, full term, normally breastfeeding infants, whose mother is willing to breastfeed during the painful procedure and consents to study participation. Normally breastfeeding infants will be defined as those infants who had fed directly at the breast a minimum of two times in the 24-hours prior to blood collection and whose mother and/or staff nurse reported active sucking and swallowing during those feeds. Infants who have undergone repeated heel lancing for blood glucose and/or bilirubin monitoring (e.g., small or large for gestational age infants, infants born to diabetic mothers, or with hyperbilirubinemia) will be considered eligible, however, diagnosis and the number of prior painful procedures will be recorded and retained for statistical analysis.

Exclusion Criteria:

* Infants will not be eligible for study participation if they are a twin birth (including all classifications of monozygotic and dizygotic twins) due to the potential for non-independence of outcomes between twin pairs, show signs of infection, significant lower limb tissue damage, have had previous surgery or intra-ventricular hemorrhage, are born to opioid using mothers or with significant genetic disorders, are unable to breastfeed or have contraindications to sucrose administration, or whose parents are unable to provide written informed consent.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Pain-specific event related potential | Isolated within the one-minute window post-procedure.
  The primary outcome measure will be pain-specific brain activity measured using a dense array neonatal electroencephalogram (EEG) recording that is time-locked to a medically required heel lance. Infant EEG activity will be recorded from a HydroCel Geodesic Sensor Net positioned according to the modified international 10/20 electrode placement system on a 128 Channel Geodesic EEG SystemTM 400 MR series (Electrical Geodesics Incorporated, Eugene, Oregon, USA). Pain-specific event related potentials will specifically be examined and isolated at electrode sites Cz, as previous research has reported pain-specific activity at this site in both infants and adults.

SECONDARY OUTCOMES:
Premature Infant Pain Profile-Revised | Baseline, 30, 60, 90, 120 seconds post-procedure.
  The PIPP-R, which has been revised from the original PIPP developed 14 years ago, is a 7-indicator composite pain measure consisting of 3 behavioural (facial actions: brow bulge, eye squeeze, and naso-labial furrow), 2 physiological (heart rate, oxygen saturation) and 2 contextual (gestational age, behavioural state) indicators of acute pain. A numerical score ranging from 0 - 3 is assigned to each indicator for a maximum score of 18 reflecting the worst possible pain in infants born at greater than 36 weeks' gestational age. A score of 6 or less is considered to indicate minimal or no pain, a score of 6 to 12 indicates mild or moderate pain, and a score of 12 or greater indicates moderate to severe pain.
Recovery | In the 30 minute window post-procedure.
  Time to recovery will be considered the amount of time in seconds that elapses until the infant's heart rate returns to baseline average values. The point at which the infant's heart rate reaches baseline levels and is sustained for no less than five to seven beats following the heel lance will indicate recovery.
Maternal acceptability | Immediately post-procedure.
  Mothers will be asked to complete an open-ended questionnaire with 3-5 questions (depending on assigned condition) following completion of the study procedures. This questionnaire will focus on assessing maternal acceptability of the use of the assigned breastfeeding or sweet taste intervention as well as the use of neurophysiological imaging technology to measure newborn pain responding in the neonatal period.

CONTACTS AND LOCATIONS:
Overall Officials: Britney L Benoit, MScN RN PhD(c), Principal Investigator — Dalhousie University & IWK Health Centre
Locations (1):
- Britney Benoit, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benoit B, Newman A, Martin-Misener R, Latimer M, Campbell-Yeo M. The influence of breastfeeding on cortical and bio-behavioural indicators of procedural pain in newborns: Findings of a randomized controlled trial. Early Hum Dev. 2021 Mar;154:105308. doi: 10.1016/j.earlhumdev.2021.105308. Epub 2021 Jan 12. PMID 33513546